CLINICAL TRIAL: NCT06238076
Title: Universal Surgical Device for Mandibular Reconstruction Using Fibula Free Flap : Feasibility Study.
Brief Title: Evaluation of an Universal Surgical Device for Mandibular Reconstruction.
Acronym: FIBUMAND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/17/0347
Record Dates: First submitted 2024-01-11; First posted 2024-02-02 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Mandibular Reconstruction
Keywords: Mandible; Mandibular Reconstruction; Computer-Aided Design; Fibular free flap; Computer Assisted three dimensional imaging; Surgical equipment

STUDY DESIGN:
Intervention Model Description: Feasibility pilot study, monocentric, non-comparative
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group experimental (Experimental): The patients included in the study and admitted in the maxillofacial surgery department for mandibular fibula free flap reconstruction will benefit from a surgery assisted with the universal surgical device FIBUMAND.
  Interventions: Device: Universal surgical device FIBUMAND

INTERVENTIONS:
Device: Universal surgical device FIBUMAND — This device is made of biocompatible resin for type IIa medical devices with a 3D printer.

SUMMARY:
Fibula free flap is the gold standard for mandibular reconstruction. The shape of the fibula requires osteotomy that can be performed with a custom surgical guide. The use of surgical guide shorten surgical time, enhances the precision of the surgeon and reduces morbidity.

Since 2008 custom surgical guide have been used in the hospital department and the clinical team have noticed a number of elements, which leads investigator to think that it would be possible to perform this kind of procedure using an universal guide.

The aim of this study is to assess the possibility to perform mandibular fibula free flap reconstruction with an universal guide.

ELIGIBILITY:
Inclusion Criteria:

* Admitted in the maxillofacial surgery department for mandibular fibula free flap reconstruction including a symphysial bone fragment
* Patients insured under the French social security system
* Free and informed consent

Exclusion Criteria:

* Lateral mandibular reconstruction without symphysis reconstruction
* Legally incompetent
* Inclusion in another protocol of research , involving mandibular reconstruction
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility of guiding mandibular fibula free flap reconstruction with an universal guide. | Day 1
  Either the surgeon assists the entire procedure using the device and the patient is registered as "success", or the device is not suitable and cannot be used and the patient is registered as " failure ". Partial use is also considered a failure of the procedure.

SECONDARY OUTCOMES:
Time of surgical procedure | Day 1
  It is timed (in minutes) during the procedure and relative to the total duration of the intervention.
Qualitative assessment of the device by the surgeon | Day 1
  Evaluation of the general appreciation according a 4-point scale (very unsatisfactory / unsatisfactory / satisfactory / excellent) about the:
  * The positioning and fixing of the guide,
  * Performing osteotomies,
  * The use of the meter,
  * The congruence of the bone surfaces,
  * The use of the plate shaper,
  * Fibular osteosynthesis,
  * The mandibular reconstruction obtained
Post-operative quality of life | From 6 to 8 weeks
  The patient's postoperative quality of life will be assessed by the University of Washington Quality of Life Questionnaire (UW-QOL) version 4.0.
  UW-QOL questionnaire consists of 12 single question domains, these having between 3 and 6 response options that are scaled evenly from 0 (worst) to 100 (best) according to the hierarchy of response. The domains are pain, appearance, activity, recreation, swallowing, chewing, speech, shoulder, taste, saliva, mood and anxiety. Another question asks patients to choose up to three of these domains that have been the most important to them. There are also three global questions, one about how patients feel relative to before they developed their cancer, one about their health-related QOL and one about their overall QOL.The whole questionnaire focuses on current patient health and quality of life within the past 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Alice PREVOST, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No